CLINICAL TRIAL: NCT03805607
Title: Prospective Evaluation of the Effects of IV Ketorolac on Platelet Function Post-Cesarean Delivery
Brief Title: IV Ketorolac on Platelet Function Post-Cesarean Delivery
Acronym: KetoPltAgg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Society for Obstetric Anesthesia and Perinatology (Other)
Responsible Party: Principal Investigator, Phillip Hess, Associate Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018P000625
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Analgesia, Obstetrical; Coagulation Defect; Postpartum; Nonsteroidals (NSAIDs)Toxicity; Postpartum Hemorrhage; Postoperative Pain; Ketorolac Adverse Reaction; Blood Loss, Postoperative
Keywords: Cesarean Section Complications; Blood Loss, Surgical; Coagulation Defect; Postpartum; Nonsteroidals (NSAIDs)Toxicity; Postpartum Hemorrhage; Ketorolac; Cesarean Delivery; Platelet Function; Cyclooxygenase Inhibitors/administration & dosage; Female; Humans; Ketorolac/administration & dosage; Pain, Postoperative/drug therapy; Pregnancy
MeSH Terms: conditions — Agnosia; Hemostatic Disorders; Postpartum Hemorrhage; Pain, Postoperative; Postoperative Hemorrhage; Blood Loss, Surgical; Pain | interventions — Ketorolac Tromethamine; Ketorolac; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized Placebo-Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo (normal saline) or ketorolac in syringe prepared by the investigational pharmacy with study patient number and blinding key maintained by investigational pharmacy until time of unblinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): 1 ml of normal saline
  Interventions: Drug: Placebos
- Ketorolac (Experimental): 30 mg of ketorolac in 1 ml
  Interventions: Drug: Ketorolac Tromethamine 30 MG/ML

INTERVENTIONS:
Drug: Ketorolac Tromethamine 30 MG/ML — Ketorolac 30 mg
  Other Names: ketorolac; Ketorolac Tromethamine; Ketorolac Injectable Solution
  Arms: Ketorolac
Drug: Placebos — Normal Saline
  Other Names: Placebo; Normal Saline
  Arms: Placebo

SUMMARY:
Cesarean delivery has become the most common surgical procedure in the US. Non-steroidal anti-inflammatory drugs (NSAIDs) have been shown to improve the quality of post-cesarean analgesia and markedly reduce opioid consumption. The effect of NSAIDs on healthy volunteers results in inhibition of platelet aggregation and prolonged bleeding time. However, in the obstetric population, the presence and degree of platelet inhibition after NSAID exposure is less clear. The investigators plan to use Platelet Aggregometry and Thromboelastography (TEG) to evaluate the effect of ketorolac on platelets.

DETAILED DESCRIPTION:
Cesarean delivery has become the most common surgical procedure in the US, with over 1.2 million cesarean deliveries performed each year. The addition of non-steroidal anti-inflammatory drugs (NSAIDs) to a post-cesarean analgesic regimen has been shown to improve the quality of post-cesarean analgesia and markedly reduce opioid consumption. As a result, fewer patients incur opioid related side-effects such as nausea and vomiting, respiratory compromise, sedation, and impaired breast-feeding.

The effect of NSAIDs on healthy volunteers is relatively well-described. Most commonly, NSAIDs inhibit membrane-bound cyclooxygenase 1 (COX-1), the enzyme responsible for the production of the platelet agonist thromboxane A2. This ultimately results in inhibition of platelet aggregation and prolonged bleeding time. However, in the obstetric population, the presence and degree of platelet inhibition after NSAID exposure is less clear. This has limited the incorporation of NSAIDs into protocols for postpartum analgesia following cesarean delivery.

Platelet Function Assessment 100 (PFA) assays, with collagen/epinephrine and collagen/ADP (adenosine diphosphate) as agonists, can reliably test for platelet inhibition. PFA has been utilized to examine the anti-platelet effects of platelet inhibitors including NSAIDs in studies involving non-obstetric patients. Similarly, platelet aggregometry has been used to evaluate the platelet inhibitory effects of NSAIDs. Thromboelastography (TEG) has been shown in numerous studies to represent in-vivo clot strength and function.

Research in this field is needed as physiologic changes of pregnancy combined with significant surgical blood loss and hemodilution at cesarean delivery may alter the effect on maternal platelet function. This has become more pressing as postpartum thromboprophylaxis is likely to be more commonly considered for patients after cesarean delivery. In their most recent unofficial guidelines, the American Society of Regional Anesthesia state that NSAIDs should not be used with thromboprophylaxis after patients received neuraxial blockade (ASRA App). However, to the best of our knowledge, there is limited data, only utilizing bleeding time,5 examining the potential platelet inhibitory effect of NSAIDs in a low-risk healthy cohort undergoing cesarean delivery.

Protocol:

Brief Study Protocol After obtaining Institutional Review Board (IRB) approval, patients will be randomly assigned to receive either IV ketorolac 30 mg (n=15) or normal saline (n=15) based on a pre-assigned randomization sequence. The assignment for each patient will be kept in sealed opaque envelopes. After obtaining written informed consent, an anesthesiologist not involved in the study will open the envelope and will prepare the study drug. The patient and the study investigators will be blinded to the study drug.

Baseline platelet count, coagulation parameters (activated partial thromboplastin time (APTT), prothrombin time (PT), Fibrinogen) and TEG parameters will be measured pre-operatively on the day of surgery. Routine lab work obtained at this time will require 10 ml of blood, while study related tests will require 5.4 ml. Each patient will undergo either spinal or combined spinal epidural anesthesia with our standard cesarean induction dose of hyperbaric intrathecal 0.75% bupivacaine 1.5 ml, intrathecal fentanyl 25 micrograms and intrathecal morphine 250 micrograms. The patient will be moved to the supine position with left lateral uterine displacement. When a T6 sensory level to pinprick is achieved, cesarean delivery will be allowed to proceed. At the completion of the surgery, Platelet Aggregometry and TEG parameters will be performed to assess for intraoperative changes to TEG and establish baseline Platelet Aggregometry values. A total volume of 18.9 ml of blood will be withdrawn for the study at this time. While under the effect of the spinal medication, meaning that the patient is unable to fill sharp in their feet, the patient may elect to have this blood and the subsequent blood drawn from their foot to avoid unnecessary pain. These blood draws would only be performed by an anesthesiologist and only if a suitable site was identified. Performing venipucture for lab draws in the feet is not known to increase the risk of complications from blood draws when compared to the upper extremity. The study drug will be administered upon completion of the case. Platelet Aggregometry and TEG parameters will be performed 10 min after study drug administration. An additional volume of 18.9 ml of blood will be withdrawn for the study at this time. After blood samples have been obtained, patients in each group will receive the alternate therapy (ie placebo group receives ketorolac and ketorolac receives placebo), allowing both groups to benefit from the analgesic effect of ketorolac. Supplemental analgesia will be administered according to a standard post-operative pain management protocol on labor and delivery.

Statistical analysis: Data will be assessed for normality using normality plots and the Kolmogorov-Smirnov test. Demographic, obstetric, and perioperative data will be presented as mean (SD) or median [interquartile range]. Between-group comparisons will be assessed using the unpaired t test and Mann-Whitney U test, where appropriate. Within-group before vs. after NSAID exposure changes will be assessed using the paired t test and Wilcoxon signed rank test, where appropriate. The percentage change from baseline for each PFA, TEG, and lab parameter will also be calculated.

Sample size justification: There is limited data on the affect of ketorolac on quantitative coagulation studies, particularly in the obstetric population. Based on available data from a prior study examining platelet inhibition of non-opioid analgesics, a PFA closure time ≥173 seconds can be used to classify platelet inhibition. Using the aforementioned data on epinephrine-induced PFA closure time, the investigators estimate that, before and after ketorolac exposure, 25% and 70% patients respectively would exhibit prolonged PFA closure times. With an alpha error of 0.05 and a beta error of 0.8, the investigators estimated that a sample size of 18 patients per group would provide 80% power. Additional studies have examined the affect of ketorolac on platelet aggregometry. Platelet aggregometry to collagen was diminished in the ketorolac group from preoperative to poststudy drug data points (90.8% +/- 7.6% to 60.5% +/- 32.5%; P < 0.01). With an alpha error of 0.05 and a beta error of 0.8, the investigators estimated that a sample size of 19 patients per group would provide 80% power.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Undergoing routine, scheduled cesarean section
* Gestation >37 weeks
* Singleton gestation
* Intraoperative anesthesia - 1.5 ml of intrathecal bupivicaine 0.75%, 25mcg of intrathecal fentanyl and 250 mcg of intrathecal morphine via Spinal or Combined Spinal Epidural

Exclusion Criteria:

* Pre-eclampsia with severe features or HELLP
* Allergy to NSAIDs
* Pre-existing bleeding disorder
* Other major risk factor for postpartum hemorrhage (placenta accreta, large uterine fibroid)
* Chronic kidney disease
* Plt count less than 100k
* Gastric ulcer or gastric bleeding
* Pre-existing uterine bleeding or disseminated intravascular coagulation
* Patient or Obstetrician refusal
* Intraoperative exclusion criteria - Postpartum hemorrhage (EBL >1000 ml) or unplanned intraoperative extension of surgery

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Platelet Aggregometry Light Transmission | 15 minutes after dosing of placebo or ketorolac
  Platelet Aggregometry uses measurements platelet rich blood or serum samples and activating agents to analyze the percent change in light transmission as a marker of platelet aggregation.

SECONDARY OUTCOMES:
Thromboelastogram parameters including Reaction time (R) | 15 minutes after dosing of placebo or ketorolac
  Thromboelastogram parameters including Reaction time (R)
Thromboelastogram parameters including Angle (alpha) | 15 minutes after dosing of placebo or ketorolac
  Thromboelastogram parameters including Angle (alpha)
Thromboelastogram parameters including Kinetics (K) | 15 minutes after dosing of placebo or ketorolac
  Thromboelastogram parameters including Kinetics (K)
Thromboelastogram parameters including Maximum Amplitude (MA) | 15 minutes after dosing of placebo or ketorolac
  Thromboelastogram parameters including Maximum Amplitude (MA)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared.

REFERENCES:
- [Background] Blackburn A, Stevens JD, Wheatley RG, Madej TH, Hunter D. Balanced analgesia with intravenous ketorolac and patient-controlled morphine following lower abdominal surgery. J Clin Anesth. 1995 Mar;7(2):103-8. doi: 10.1016/0952-8180(94)00040-b. PMID 7598916
- [Background] Diemunsch P, Alt M, Diemunsch AM, Treisser A. Post cesarean analgesia with ketorolac tromethamine and uterine atonia. Eur J Obstet Gynecol Reprod Biol. 1997 Apr;72(2):205-6. doi: 10.1016/s0301-2115(96)02682-6. No abstract available. PMID 9134403
- [Background] Pavy TJ, Paech MJ, Evans SF. The effect of intravenous ketorolac on opioid requirement and pain after cesarean delivery. Anesth Analg. 2001 Apr;92(4):1010-4. doi: 10.1097/00000539-200104000-00038. PMID 11273941
- [Background] Lowder JL, Shackelford DP, Holbert D, Beste TM. A randomized, controlled trial to compare ketorolac tromethamine versus placebo after cesarean section to reduce pain and narcotic usage. Am J Obstet Gynecol. 2003 Dec;189(6):1559-62; discussion 1562. doi: 10.1016/j.ajog.2003.08.014. PMID 14710063
- [Background] El-Tahan MR, Warda OM, Yasseen AM, Attallah MM, Matter MK. A randomized study of the effects of preoperative ketorolac on general anaesthesia for caesarean section. Int J Obstet Anesth. 2007 Jul;16(3):214-20. doi: 10.1016/j.ijoa.2007.01.012. Epub 2007 Apr 24. PMID 17459695
- [Background] Elhakim M, Fathy A, Amine H, Saeed A, Mekawy M. Effect of i.v. tenoxicam during caesarean delivery on platelet activity. Acta Anaesthesiol Scand. 2000 May;44(5):555-9. doi: 10.1034/j.1399-6576.2000.00512.x. PMID 10786742
- [Background] Gobble RM, Hoang HLT, Kachniarz B, Orgill DP. Ketorolac does not increase perioperative bleeding: a meta-analysis of randomized controlled trials. Plast Reconstr Surg. 2014 Mar;133(3):741-755. doi: 10.1097/01.prs.0000438459.60474.b5. PMID 24572864